CLINICAL TRIAL: NCT06303531
Title: An Interventional, Single-Center, Randomized, Unblinded, Parallel-Group, Three-Arm Study to Investigate the Superiority of 12 Weeks of Oral Treatment With Ferrous Ascorbate (EBMfer) or Ferrous Fumarate (Eurofer) as Compared to Polysaccharide Iron (FeraMAX) in Hemoglobin Level Changes in Adults Aged 18 and Above With Iron Deficiency Anemia (EFFICACIOUS IRON)
Brief Title: Efficacious Iron for Iron Deficiency Anemia in Adults Aged ≥18 Years
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Anil K. Gupta Medicine Professional Corporation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Efficacious Iron
Record Dates: First submitted 2024-02-26; First posted 2024-03-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Anemia; Iron Deficiency; Ferrous Fumarate; Polysaccharide Iron; Ferrous Ascorbate
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies | interventions — ferrous fumarate; Niferex; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eurofer (Active Comparator): Ferrous Fumarate - 300 mg
  Interventions: Dietary Supplement: Ferrous Fumarate
- FeraMAX (Active Comparator): Polysaccharide Iron - 150mg
  Interventions: Dietary Supplement: Polysaccharide Iron
- EBMfer (Active Comparator): Ferrous Ascorbate - 100 mg
  Interventions: Dietary Supplement: Ferrous Ascorbate

INTERVENTIONS:
Dietary Supplement: Ferrous Fumarate — Ferrous Fumarate - 300 mg
  Other Names: Eurofer
  Arms: Eurofer
Dietary Supplement: Polysaccharide Iron — Polysaccharide Iron - 150 mg
  Other Names: FeraMAX
  Arms: FeraMAX
Dietary Supplement: Ferrous Ascorbate — Ferrous Ascorbate - 100 mg
  Other Names: EBMfer
  Arms: EBMfer

SUMMARY:
Iron deficiency anemia (IDA) is a widespread condition affecting many people globally. Despite the many cases of IDA, there are few studies that compare the effectiveness of different types of iron supplements with a greater emphasis on the cost of supplements and their tolerability. This study aims to conduct a comparison between different iron supplements to determine the superiority of the iron supplements Ferrous Ascorbate (EBMfer) and Ferrous Fumarate (Eurofer) over polysaccharide iron (FeraMax). This comparison will be conducted by determining the change in hemoglobin levels for participants in this trial over a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥18 years of age when signing the informed consent.
2. Participants with iron deficiency anemia are defined as follows for the purpose of this study:

Male: Hgb > 80 to ≤135g/L and Serum Ferritin < 30 ug/L Female: Hgb > 80 to ≤120g/L and Serum Ferritin < 30 ug/L 2b. Local lab done prior to 7 days can be enrolled in the trial provided all the inclusion and exclusion criteria are met.

2c. Previously Screen Failed subjects not meeting the <15 ug/L ferritin criteria can be rescreened once ICF is signed.

2d. Subjects not on iron supplement and meeting all the randomization criteria do not have to wait for 7 days for visit 2.

3. Sex and Contraceptive/Barrier Requirements, Male and Female participants: None 4. Must have given written informed consent (signed and dated) 5. Medication Stopping: If the participant is currently on an iron supplement, they must be willing to discontinue the medication upon signing the Informed Consent Form (ICF) and throughout the study. 6. Protocol Compliance: Participants must be able to comply with the requirements outlined in the study protocol

Exclusion Criteria:

1. Hemoglobin (Hb) ≤ 80 g/L
2. Medical history of current hematological disorders other than iron deficiency anemia (e.g., aplastic anemia, megaloblastic anemia, sideroblastic anemia, pernicious anemia, thalassemia trait, thalassemia, sickle cell anemia, etc.).
3. Medical history of chronic renal disease, current history of any known inflammatory disorder, and any chronic medical condition that, in the opinion of the Principal Investigator, would compromise participant safety.
4. Medical history or evidence of intestinal malabsorption, malabsorption syndrome, hemochromatosis, and hemosiderosis, hypochlorhydria, achlorhydria, gastrectomy, and gastrojejunostomy.
5. History of occult blood in the stool.
6. Obvious internal or external bleeding as documented by medical history if considered clinically significant in the investigator's opinion.
7. Severe and uncontrolled diseases, including serious psychological disorders, that are likely to interfere with the study.
8. Significant co-morbidity, such as a severe chronic medical condition unrelated to iron deficiency that is apparent on history or laboratory tests.
9. Iron Supplementation: Throughout the study duration, participants are not allowed to receive other sources of iron supplementation, including but not limited to other oral iron tablets and intravenous iron therapy.
10. Prohibited Medication: Inability to withhold prohibited medications. Prohibited medications include Proton Pump Inhibitors, Cholestyramine, colestipol, and new anticoagulant therapy initiated in the past six months (e.g., warfarin, apixaban, dabigatran, edoxaban, rivaroxaban).
11. Multivitamin and Mineral Supplements: Not willing to discontinue multivitamin and mineral supplements containing 35 mg or more of elemental iron per day on the day of screening and throughout the study.
12. Blood Transfusion, Blood Donation, and IV Iron Therapy: History of blood transfusion, blood donation, or significant blood loss (e.g., due to an accident or surgery), or intravenous iron therapy in the past four months.
13. Participants must not be currently participating in any other interventional clinical trial.
14. Pregnancy: A urine dipstick pregnancy test will be performed at Visit 1, and pregnant individuals will be excluded from the study.
15. Desire to Conceive Within the Next 13 weeks: This criterion includes patients who are actively trying to conceive or are receiving treatment to facilitate conception. They will be excluded from the study.
16. Known or Suspected Hypersensitivity to Iron: Individuals with a known or suspected hypersensitivity to iron or any of the components of Ferrous Fumarate (Eurofer), Polysaccharide Iron (FeraMAX), and Ferrous Ascorbate (EBMfer) will be excluded.
17. Planned Surgery: Participants with planned surgery during the study or those who had surgery within two weeks before the screening visit will be excluded.
18. Difficulties with Blood Sampling: Individuals with difficulties related to blood sampling that might hinder the study procedures will be excluded.
19. Alcohol or Drug Abuse: Participants showing evidence of alcohol or drug abuse that, in the opinion of the investigator, could interfere with study compliance or prevent understanding of the study's objectives and procedures will be excluded.
20. Inability to Follow Study Procedures: This includes individuals who are unable to follow study procedures due to factors like language problems or self-reported psychological disorders.
21. Enrollment of the Investigator, Family Members, and Clinic Employees: The investigator, their family members, and clinic employees will not be eligible to participate in the study to avoid any potential conflicts of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin Levels | 12 Weeks from Baseline
  Hemoglobin levels measured using a hematology panel at baseline and 12 weeks

SECONDARY OUTCOMES:
Change in Serum Ferritin | 12 Weeks from Baseline
  Serum ferritin measured using a hematology panel at baseline and 12 weeks
Tolerability of Study Medication - Discontinuation Rate | 12 Weeks from Baseline
  Discontinuation rates measured using subject compliance over the trial period of 12 weeks. Discontinuation rate will be measured based on subject compliance with study medication as a rate based on time.

CONTACTS AND LOCATIONS:
Locations (1):
- Albion Finch Medical Centre, Etobicoke, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ganguly S. Comparison between Ferrous Ascorbate and Colloidal Iron in the Treatment of Iron Deficiency Anemia in Children from Kolkata, India. BJMMR 2012; 2: 195-205.
- [Background] Powers JM, Buchanan GR, Adix L, Zhang S, Gao A, McCavit TL. Effect of Low-Dose Ferrous Sulfate vs Iron Polysaccharide Complex on Hemoglobin Concentration in Young Children With Nutritional Iron-Deficiency Anemia: A Randomized Clinical Trial. JAMA. 2017 Jun 13;317(22):2297-2304. doi: 10.1001/jama.2017.6846. PMID 28609534
- [Background] Liu TC, Lin SF, Chang CS, Yang WC, Chen TP. Comparison of a combination ferrous fumarate product and a polysaccharide iron complex as oral treatments of iron deficiency anemia: a Taiwanese study. Int J Hematol. 2004 Dec;80(5):416-20. doi: 10.1532/ijh97.a10409. PMID 15646652
- [Background] Moe S, Grill AK, Allan GM. Newer iron supplements for anemia. Can Fam Physician. 2019 Aug;65(8):556. No abstract available. PMID 31413026